CLINICAL TRIAL: NCT01763645
Title: International Multicenter Randomized Double Blind Phase III Trial Comparing Safety and Efficacy of BCD-021 (CJSC BIOCAD, Russia) and Paclitaxel + Carboplatin to Avastin® (F. Hoffmann-La Roche Ltd, Switzerland) and Paclitaxel + Carboplatin in Inoperable or Advanced Non-squamous Non-small-cell Lung Cancer (NSCLC) Patients
Brief Title: A Safety and Efficacy Study of BCD-021 With Paclitaxel and Carboplatin Compared to Avastin With Paclitaxel and Carboplatin in Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-021-02
Record Dates: First submitted 2012-12-27; First posted 2013-01-09 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2023-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; bevacizumab; pharmacokinetics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-021 (CISC BIOCAD) (Experimental): BCD-021 is a product code for bevacizumab biosimilar manufactured by CJSC BIOCAD, Russia. In this arm patients will receive 6 courses of treatment with BCD-021 in combination with carboplatin and paclitaxel. BCD-021 will be administered at a dose of 15 mg/kg as 90 min intravenous infusion every 3 weeks (on Day 1 of each course). Paclitaxel will be administered at a dose of 175 mg/m2 as 3 hour intravenous infusion every 3 weeks on Day 1 and carboplatin (AUC 6 mg/ml×min) as 15 - 30 min intravenous infusion just after paclitaxel every 3 weeks on Day 1.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin
- Avastin (F. Hoffmann-La Roche Ltd) (Active Comparator): In this arm patients will receive 6 courses of treatment with Avastin in combination with carboplatin and paclitaxel. Avastin will be administered at a dose of 15 mg/kg as 90 min intravenous infusion every 3 weeks on Day 1. Paclitaxel will be administered at a dose of 175 mg/m2 as 3 hour intravenous infusion every 3 weeks on Day 1 and carboplatin (AUC 6 mg/ml×min) as 15 - 30 min intravenous infusion just after paclitaxel every 3 weeks on Day 1.
  Interventions: Drug: Bevacizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Bevacizumab — Patients will receive 6 courses of bevacizumab in combination with carboplatin and paclitaxel. Bevacizumab will be administered at a dose of 15 mg/kg as 90 min intravenous infusion every 3 weeks (on Day 1 of each cycle).
  Other Names: Avastin; BCD-021
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 175 mg/m2 as 3 hour intravenous infusion on Day 1 of each 3-week course (6 courses totally)
  Other Names: Taxacad
Drug: Carboplatin — Carboplatin will be administered (AUC 6 mg/ml×min) as 15 - 30 min intravenous infusion just after paclitaxel on Day 1 of each 3-week course (6 courses totally).

SUMMARY:
BCD-021-02 is a double-blind randomized clinical trial comparing efficacy of BCD-021 (INN: bevacizumab) and paclitaxel + carboplatin to Avastin and paclitaxel + carboplatin in inoperable or advanced non-squamous NSCLC patients with pharmacokinetics substudy. The purpose of the study is to demonstrate the non-inferiority of efficacy and safety of BCD-021 compared to Avastin. Also study includes pharmacokinetics assessment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Newly diagnosed histologically or cytologically confirmed NSCLC excluding squamous NSCLC (mixed cancer types should be classified according to the prevalent cell type);
* IIIb or IV stage of NSCLC (TNM classification version 6);
* Age ≥ 18 years and age ≤ 75 years (both inclusive);
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2, (not declining within 2 weeks prior to the first dose of investigational product);
* Life expectancy - 12 weeks or more from the moment of randomization;
* Presence of at least 1 measurable tumour with a size not less than 1 cm (revealed with CT slice thickness not more than 5 mm), as defined by modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria (specifically, no ascites, pleural, or pericardial effusions, osteoblastic bone metastases, or carcinomatous lymphangitis of the lung as only lesion;
* Patients should be able to follow the Protocol procedures (according to Investigator's assessment);
* Patients must implement reliable contraceptive measures during all the study treatment, starting 4 weeks prior to the administration of the first dose of investigational product until 6 months after the last dose of investigational product. This requirement does not apply to participants who have undergone surgical sterilization, or patients who are postmenopausal (documented) for the past 2 years. Reliable contraceptive measures include two methods of contraception, including one barrier method

Exclusion Criteria:

* Squamous NSCLC;
* Proven coagulopathy, clinically significant hemorrhage in the past including nasal hemorrhage;
* absolute neutrophil count <1500/mm3;
* Platelets <100 000/mm3;
* Hemoglobin < 90 g/L;
* Creatinine level ≥1.5 mg/dL;
* Bilirubin level ≥1.5 × upper limit of normal (ULN);
* Aspartate-aminotransferase(AST) and alanine-aminotransferase (ALT) levels ≥2.5 × ULN (≥5 × ULN for patients with liver metastases);
* Alkaline phosphatase level ≥5 × ULN;
* Current therapeutic anticoagulation treatment, aspirin (more than 325 mg/day), nonsteroidal anti-inflammatory drugs, antiplatelet agents or protracted treatment with these drugs less than 1 month before entering the study;
* Uncontrolled hypertension comprising all cases of arterial hypertension when no decrease in blood pressure could be achieved despite treatment with a combination of 3 antihypertensive drugs including one diuretic and non-medical correction methods (low salt diet, physical exercise);
* Any previous anticancer therapy (chemotherapy, radiation therapy , surgery etc.) of metastatic NSCLC;
* Radiation or hormone therapy within 21 days prior to randomization;
* Major surgery 28 days before inclusion into the study;
* Previous antiangiogenic therapy;
* Hypersensitivity to taxanes, platinum agents, recombinant murine proteins, contrast agents, premedication agents specified by Protocol (dexamethasone, diphenhydramine, ranitidine) or excipients of investigational products;
* NSCLC metastases in central nervous system excluding metastases non-progressing without glucocorticosteroids within 4 weeks before inclusion into the trial;
* Cardiovascular system pathology (CHF stage III-IV according to New York Heart Association (NYHA) classification);
* Pregnancy or lactation;
* Conditions limiting patient's adherence to Protocol requirements (dementia, neurologic or psychiatric disorders, drug addiction, alcoholism and others);
* Stage II-IV neuropathy according to Common Terminology Criteria for Adverse Events (CTCAE) v.4.0;
* Simultaneous participation in other clinical trials, previous participation in other clinical trials within 30 days before entering into the trial, previous participation in the same trial;
* Any other concomitant cancer revealed within 5 years prior to screening, except curatively treated intraductal carcinoma in situ, curatively treated cervical carcinoma in situ or curatively treated basal cell or squamous cell carcinoma;
* Acute or active chronic infections;
* Hepatitis C virus, hepatitis B virus, HIV, or syphilis infections;
* Obstacles in intravenous administration of study drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Linkova, MD, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (44):
- Belarus (4):
  - Brest Regional Clinical Dispensary, Brest
  - Grodno Regional Clinical Hospital, Grodno
  - Gomel Regional Clinical Oncology Dispensary, Homyel
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- India (3):
  - HCG Bangalore Institute of Oncology, Bangalore
  - M.S.Ramaiah Memorial Hospital, Bangalore
  - Narayana Hrudayalaya Hospitals, Bangalore
- Russia (27):
  - Arkhangelsk District Clinical Oncology Dispensary, Arkhangelsk
  - Non-governmental Healthcare Institution "Railway Clinical hospital on the Chelyabinsk Station of JSC Russian Railways", Chelyabinsk
  - State-financed Health Institution "Chelyabinsk Region Clinical Oncology Dispansary", Chelyabinsk
  - State Healthcare Facility "Kursk Regional Oncology Dispensary", Kursk
  - Institution of Russian Academy of Medical Sciences "Russian Cancer Research Center named after N.N. Blokhin", Moscow
  - Federal State Institution "Moscow Institute of Cancer Research named after P.A. Hertsen" Ministry of Health of Russian Federation, Moscow
  - State Health Institution of Moscow "Moscow City Oncology Hospital #62 of Moscow Board of Health", Moscow Region
  - Murmansk Regional Oncology Dispensary, Murmansk
  - Nizhny Novgorod Region State Budgetary Healthcare Facility "Clinical Diagnostics Center", Nizhny Novgorod
  - State Healthcare Facility "Nizhny Novgorod Regional Oncology Dispensary", Nizhny Novgorod
  - City Clinical Hospital №1, Novosibirsk
  - Regional State Health Institution "Orlov Oncology Dispansary", Oryol
  - State Health Institution "Region Oncology Dispansary", Penza
  - Perm Region Oncology Dispensary, Perm
  - Federal Government Budgetary Institution "Rostov Institute of Cancer Research" of Ministry of Health of Russian Federation, Rostov-on-Don
  - Saint Petersburg City Clinical Oncology Center, Saint Petersburg
  - St. Petersburg State Medical University n.a. I. P. Pavlov, Saint Petersburg
  - N.N.Petrov Oncology Research Center, Saint Petersburg
  - St. Petersburg Research and Practice Center for Secondary Care in Oncology, Saint Petersburg
  - Military Medical Academy named after S.M. Kirov, Saint Petersburg
  - Russian scientific center of radiology and surgery technologies, Saint Petersburg
  - State-financed Health Institution "Samara Region Clinical Oncology Dispansary", Samara
  - Oncology Dispensary 2, Sochi
  - State-financed Health Institution "Stavropol Region Clinical Oncology Dispansary", Stavropol
  - Volgograd District Oncology Dispensary №1, Volgograd
  - Volgograd Regional Oncology Dispensary №3, Volgograd
  - State Health Institution "Voronezh Region Clinical Oncology Dispansary", Voronezh
- Ukraine (10):
  - Donetsk City Oncology Dispensary, Donetsk
  - Donetsk Regional Antitumor Center, Donetsk
  - Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Kryvyi Rih Oncology Dispensary, Kryvyi Rih
  - Lviv State Regional Cancer Diagnostic and Treatment Center, Lviv
  - City Hospital № 2, Makiivka
  - Poltava Regional Clinical Oncology Dispensary, Poltava
  - Zakarpatskyi Clinical Oncology Dispensary, Uzhhorod
  - Vinnytsia Regional Clinical Oncology Dispensary, Vinnytsia
  - Zaporizhia Regional Clinical Oncology Dispensary, Zaporizhia

REFERENCES:
- [Derived] Stroyakovskiy DL, Fadeeva NV, Matrosova MP, Shelepen KG, Adamchuk GA, Roy B, Nagarkar R, Kalloli M, Zhuravleva D, Voevodin GD, Shustova MS, Kryukov F. Randomized double-blind clinical trial comparing safety and efficacy of the biosimilar BCD-021 with reference bevacizumab. BMC Cancer. 2022 Feb 1;22(1):129. doi: 10.1186/s12885-022-09243-7. PMID 35105329
- See also: Stroyakovskiy, D.L., Fadeeva, N.V., Matrosova, M.P. et al. Randomized double-blind clinical trial comparing safety and efficacy of the biosimilar BCD-021 with reference bevacizumab. BMC Cancer 22, 129 (2022). https://doi.org/10.1186/s12885-022-09243-7 — https://doi.org/10.1186/s12885-022-09243-7

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 343 of 353 patients received at least one dose of the study drug/comparator. 10 patients discontinued the study without receiving a single dose of the study drug/comparator. The safety analysis included all data from all randomized subjects who received at least one dose of study therapy, 2 of 343 patients were excluded from the efficacy analysis due to screening failure (1 in each group), n= 341.
Groups:
- BCD-021 (CISC BIOCAD): In this arm patients received 6 courses of treatment with BCD-021 in combination with carboplatin and paclitaxel. BCD-021 was administered at a dose of 15 mg/kg as 90 min intravenous infusion every 3 weeks (on Day 1 of each course). Paclitaxel was administered at a dose of 175 mg/m2 as 3 hour intravenous infusion every 3 weeks on Day 1 and carboplatin (AUC 6 mg/ml×min) as 15 - 30 min intravenous infusion just after paclitaxel every 3 weeks on Day 1.
- Avastin (F. Hoffmann-La Roche Ltd): In this arm patients received 6 courses of treatment with Avastin in combination with carboplatin and paclitaxel. Avastin was administered at a dose of 15 mg/kg as 90 min intravenous infusion every 3 weeks on Day 1. Paclitaxel was administered at a dose of 175 mg/m2 as 3 hour intravenous infusion every 3 weeks on Day 1 and carboplatin (AUC 6 mg/ml×min) as 15 - 30 min intravenous infusion just after paclitaxel every 3 weeks on Day 1.
Period: Overall Study
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
Started | 211 | 142
Received at Least 1 Dose of Study Drug | 206 | 137
Completed | 87 (Completed the study according the protocol.) | 56 (Completed the study according the protocol.)
Not Completed | 124 | 86

BASELINE CHARACTERISTICS:
Population: Patients who received at least 1 dose of the study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd) | Total
Number analyzed (Participants) | 206 | 137 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.79 (8.88) | 58.67 (8.33) | 58.23 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 of 343 participants were excluded from the analysis due to screening failure (1 in each group). 341 participants were analyzed (205 participants in BCD-021 group and 136 participants in Avastin group)
  Participants
    number analyzed (Participants) | 205 | 136 | 341
    Female | 142 | 88 | 230
    Male | 63 | 48 | 111

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Day 127
Population: The efficacy analysis included only those patients who received at least one dose of BCD-021 or Avastin®, and in whom it was possible to assess the response to therapy.
Measure: Number; unit: percentage of participans
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
Number analyzed (Participants) | 163 | 107
percentage of participans | 34.63 | 33.82

2. Primary Outcome: Area Under the Curve After the First Test Drug Administration
Description: primary outcome measure for pharmacokinetics (PK) substudy
Time Frame: up to Day 22, after the first bevacizumab administration (time points for blood samples: 0 h 1.5 h, 3 h, 4.5 h, 6 h, 24 h, 96 h, 168 h, 336 h and 504 h)
Population: Patients who received one dose of study drug and after 504 hours after injection had missed <= 1 blood sample collection to analyze pharmacokinetics.
Measure: Median (Full Range); unit: (ng/ml)*hour
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
Number analyzed (Participants) | 111 | 58
(ng/ml)*hour | 26951463 [6114172.35 to 68355846] | 23970112.875 [8216733.75 to 80859445.5]

3. Secondary Outcome: Complete Response Rate
Description: secondary outcome measure for efficacy evaluation
Time Frame: Day 127
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
Number analyzed (Participants) | 54 | 56
percentage of patients | 1.85 [0.33 to 9.77] | 1.79 [0.32 to 9.45]

4. Secondary Outcome: Partial Response Rate
Description: secondary outcome measure for efficacy evaluation
Time Frame: Day 127
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
Number analyzed (Participants) | 54 | 56
percentage of patients | 40.74 [28.68 to 54.03] | 37.50 [26.01 to 50.59]

5. Secondary Outcome: Stabilization Rate
Description: secondary outcome measure for efficacy evaluation
Time Frame: Day 127
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
Number analyzed (Participants) | 54 | 56
percentage of patients | 51.85 [38.85 to 64.60] | 51.79 [39.01 to 64.34]

6. Secondary Outcome: Progression Rate
Description: secondary outcome measure for efficacy evaluation
Time Frame: Day 127
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
Number analyzed (Participants) | 54 | 56
percentage of patients | 5.56 [1.91 to 15.11] | 8.93 [3.88 to 19.26]

7. Secondary Outcome: Occurrence of Anti-bevacizumab Antibodies
Description: Secondary outcome measure for immunogenicity assessment
Time Frame: Day 1 (before the drug administration), Day 15, 64 and 127
Measure: Number; unit: percentage of patients
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
Number analyzed (Participants) | 68 | 66
percentage of patients | 1.47 | 1.52

ADVERSE EVENTS:
Time Frame: 6 therapy cycles
Description: The safety analysis included all subjects who received at least one dose of BCD-021 or Avastin® (n = 343).
Groups:
- BCD-021 (CISC BIOCAD): In this arm patients received 6 courses of treatment with BCD-021 in combination with carboplatin and paclitaxel. BCD-021 was administered at a dose of 15 mg/kg as 90 min intravenous infusion every 3 weeks (on Day 1 of each course). Paclitaxel was administered at a dose of 175 mg/m2 as 3 hour intravenous infusion every 3 weeks on Day 1 and carboplatin (AUC 6 mg/ml×min) as 15 - 30 min intravenous infusion just after paclitaxel every 3 weeks on Day 1.
  Data on adverse events was collected from date of signing informed consent up to 18 weeks after first injection of study drug.
- Avastin (F. Hoffmann-La Roche Ltd): In this arm patients received 6 courses of treatment with Avastin in combination with carboplatin and paclitaxel. Avastin was administered at a dose of 15 mg/kg as 90 min intravenous infusion every 3 weeks on Day 1.
  Paclitaxel was administered at a dose of 175 mg/m2 as 3 hour intravenous infusion every 3 weeks on Day 1 and carboplatin (AUC 6 mg/ml×min) as 15 - 30 min intravenous infusion just after paclitaxel every 3 weeks on Day 1.
  Data on adverse events was collected from date of signing informed consent up to 18 weeks after first injection of study drug.
Arm/Group | BCD-021 (CISC BIOCAD) | Avastin (F. Hoffmann-La Roche Ltd)
All-Cause Mortality (participants affected / at risk) | 14/206 | 8/137
Serious Adverse Events (participants affected / at risk) | 36/206 | 20/137
Other Adverse Events (participants affected / at risk) | 206/206 | 137/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-021 (CISC BIOCAD) (N=206) | Avastin (F. Hoffmann-La Roche Ltd) (N=137)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Fournier's gangrene (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 2 (2)
Disease progression (General disorders) | 3 (3) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCD-021 (CISC BIOCAD) (N=206) | Avastin (F. Hoffmann-La Roche Ltd) (N=137)
Anaemia (Blood and lymphatic system disorders) | 104 (104) | 78 (78)
Thrombocytopenia (Blood and lymphatic system disorders) | 60 (60) | 42 (42)
Neutropenia (Blood and lymphatic system disorders) | 45 (45) | 37 (37)
Leukopenia (Blood and lymphatic system disorders) | 42 (42) | 39 (39)
Leukocytosis (Blood and lymphatic system disorders) | 25 (25) | 25 (25)
Neutrophilia (Blood and lymphatic system disorders) | 19 (19) | 27 (27)
Lymphopenia (Blood and lymphatic system disorders) | 23 (23) | 18 (18)
Erythropenia (Blood and lymphatic system disorders) | 17 (17) | 15 (15)
Thrombocytosis (Blood and lymphatic system disorders) | 14 (14) | 17 (17)
Lymphocytosis (Blood and lymphatic system disorders) | 13 (13) | 16 (16)
Polycythaemia (Blood and lymphatic system disorders) | 10 (10) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 25 (25) | 20 (20)
Blood alkaline phosphatase increased (Investigations) | 22 (22) | 18 (18)
Alanine aminotransferase increased (Investigations) | 19 (19) | 17 (17)
Aspartate aminotransferase increased (Investigations) | 17 (17) | 14 (14)
Blood uric acid increased (Investigations) | 18 (18) | 12 (12)
White blood cell count decreased (Investigations) | 20 (20) | 9 (9)
Blood creatinine increased (Investigations) | 12 (12) | 11 (11)
Blood pressure systolic increased (Investigations) | 12 (12) | 5 (5)
Blood urea increased (Investigations) | 6 (6) | 11 (11)
Asthenia (General disorders) | 26 (26) | 17 (17)
Pyrexia (General disorders) | 23 (23) | 14 (14)
Pain (General disorders) | 16 (16) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 53 (53) | 27 (27)
Hyperglycaemia (Metabolism and nutrition disorders) | 39 (39) | 34 (34)
Diarrhoea (Gastrointestinal disorders) | 22 (22) | 10 (10)
Nausea (Gastrointestinal disorders) | 13 (13) | 9 (9)
Neuropathy peripheral (Nervous system disorders) | 23 (23) | 16 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7)
Hypertension (Vascular disorders) | 20 (20) | 9 (9)
Tachycardia (Cardiac disorders) | 14 (14) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No